CLINICAL TRIAL: NCT03643315
Title: Determinants of Post-Exercise Eating Patterns / Alternative Title (Cover): Effect of Pre-meal Activities on Blood Pressure in Healthy Adults
Brief Title: Determinants of Post-Exercise Eating Patterns
Acronym: DEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Aaron Sim, Research Fellow, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2017/01034
Record Dates: First submitted 2018-08-07; First posted 2018-08-22 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: Appetite regulation; Eating behaviour; Exercise; HIIT
MeSH Terms: conditions — Obesity; Feeding Behavior; Motor Activity | interventions — Exercise; Meals

STUDY DESIGN:
Intervention Model Description: The present study will be of a randomised counterbalanced repeated-measures (crossover) design. Each participant (n = 30) will complete four sessions; one initial screening session (remotely administered), one baseline/familiarisation session (first lab visit) and two subsequent experimental sessions (second and third lab visits). The two experimental sessions will follow a similar protocol, except that one condition will involve an exercise protocol before an ad-libitum meal (Exercise and Meal (EX) condition), and the other, a no-exercise period (rest) before an ad-libitum (NEX) control condition.
Who Masked: Participant
Masking Description: Participants are "blind" to the true aim of the study. In addition, assignment of the experimental sessions are administered at random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Meal (EX) (Experimental): The EX protocol will involve a 30 minute acute bout of high intensity intermittent exercise on a stationary exercise bike followed by an ad-libitum test meal.
  Interventions: Behavioral: Exercise and Meal (EX)
- No-Exercise and Meal (NEX) (Experimental): The NEX protocol will involve a 30 minute period of rest (to match the exercise period in EX) where participants will be provided a video/movie. Following this, participants will be provided ad-libitum access to a test meal (as per EX energy intake assessment protocol)
  Interventions: Behavioral: No-Exercise and Meal (NEX)

INTERVENTIONS:
Behavioral: Exercise and Meal (EX) — 30 minute acute bout of high intensity intermittent exercise followed by ad-libitum meal
  Arms: Exercise and Meal (EX)
Behavioral: No-Exercise and Meal (NEX) — 30 minute non-exercise period where participants will be watching a video/movie followed by ad-libitum meal
  Arms: No-Exercise and Meal (NEX)

SUMMARY:
This study examines potential physiological and psychological determinants of food intake in response to exercise. Specifically, beyond measuring actual food consumption and physiological markers typically assessed during exercise and appetite work (i.e. appetite hormones, blood glucose), the investigators wish to investigate the influence of individual behavioural differences (attitudes towards eating, licensing/compensatory health beliefs, self-regulation, and exercise-associated motivation) on the relationship between exercise and eating behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Inactive (< 90 min of moderate-intensity exercise a week)
* BMI: 23 and above
* Age between 21 to 40 years
* Normal fasting blood glucose levels equal to or less than 5.9 mmol/L
* Non-smoker
* No know allergies or intolerance to food
* Not on any prescribed medication
* No physical disabilities and/or restrictions; not averse to exercising on a stationary bike or treadmill running
* No aversion to blood sampling procedures (e.g. finger prick, cannulation)

Exclusion Criteria:

* Female,
* Smoker,
* Fasting blood glucose > 5.9 mmol/L,
* Resting blood pressure > 140/90 mmHg,
* Any major medical/health conditions including

  * Diabetes,
  * Metabolic disease
  * Hypertension,
  * Cardiovascular disease,
  * Thyroid disorders,
  * G6PD deficiency.
* Allergic or intolerant to foods presented in the study.
* Physical disabilities and/or restrictions.
* Individuals that are adverse to exercising on a stationary exercise bike or treadmill.
* Adverse to blood sampling procedures (i.e. cannulation, finger pricks, venepuncture).

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Ad-libitum amount of food consumed in response to experimental condition: exercise or rest (no exercise). | 3 hours
  Participants' eating behaviour will be assessed by measuring the total amount of the test meal consumed in each experimental condition. The test meal will be provided ad-libitum (i.e. there will be non-restricted access)

SECONDARY OUTCOMES:
Appetite-related blood hormone concentration in response to experimental conditions. | 3 hours
  Venous blood will be sampled for the measurement of a range of appetite-related hormones including Active Ghrelin (pg/ml), Glucagon-like Peptide-1 (GLP-1) (pg/ml), Pancreatic YY (PYY) (pg/ml), Pancreatic Polypeptide (PP) (pg/ml), periodically through the experimental sessions.
Metabolic blood variable concentration in response to experimental conditions | 3 hours
  Venous blood will be sampled for the measurement of metabolic blood variables blood insulin (mmol/L) and blood glucose (mmol/L) periodically through the experimental sessions.
Subjective ratings of hunger in response to experimental conditions | 3 hours
  Self-reported subjective ratings of hunger will be assessed periodically through the experimental session. Assessed via 100-point visual analogue scales.
Subjective ratings of satiation (fullness) in response to experimental conditions | 3 hours
  Self-reported subjective ratings of satiation (fullness) will be assessed periodically through the experimental session. Assessed via 100-point visual analogue scales
Subjective ratings of desire to eat in response to experimental conditions | 3 hours
  Self-reported subjective ratings of desire to eat will be assessed periodically through the experimental session. Assessed via 100-point visual analogue scales
Subjective ratings of prospective food consumption in response to experimental conditions | 3 hours
  Self-reported subjective ratings of prospective food consumption will be assessed periodically through the experimental session. Assessed via 100-point visual analogue scales.
Free-living energy intake (1 day post-experiment) in response to experimental conditions | 1 day
  1 day free-living energy intake (self-report)
Free-living physical activity levels intake (1 day post-experiment) in response to experimental conditions | 1 day
  1 day free-living physical activity levels (physical activity monitors)

OTHER OUTCOMES:
Self-reported tendencies of compensatory health beliefs | Assessed at start of study - through study completion - up to 4-5 weeks
  Influence of self-reported tendencies of compensatory health beliefs on the relationship between experimental conditions and study outcomes. Scale to be used:
  Compensatory Health Belief (CHB) Scale, CHB Subscales: Substance use, Eating/sleeping habits, Stress and Weight regulation, Ratings on a 5-point agreement scale. Greater scores (summed) indicate greater tendency for an individual to hold compensatory beliefs (for the particular domain/subscale or collectively).
Self-reported tendencies of licensing/reward beliefs | Assessed at start of study - through study completion - up to 4-5 weeks
  Influence of self-reported tendencies of licensing eating behaviour in response to exercise on the relationship between experimental conditions and study outcomes. Scale to be used:
  Post-Exercise Licensing (PEL)Scale. Ratings on a 7 point agreement scale. Greater scores (averaged) indicate a greater tendency to reward/license in response to exercise.
Self-reported tendencies and motives of compensatory eating behaviour in response to exercise | Assessed at start of study - through study completion - up to 4-5 weeks
  Influence of self-reported tendencies and motives of compensatory eating behaviour in response to exercise on the relationship between experimental conditions and study outcomes Scale to be used:
  Compensatory Eating Motives Questionnaire (CEMQ) Subscales: Eating for Reward, Eating for Recovery, Eating for Relief (4 point frequency scale) Greater scores (summation of outcome of respective subscales) indicate greater tendency to compensate due to particular motive (respective subscales).
Self-reported assessment of motivation (regulation) to exercise | Assessed at start of study - through study completion - up to 4-5 weeks
  To examine the influence of self-reported motivation to exercise on the relationship between experimental conditions and study outcomes. Scale involve:
  Behavioural Regulation in Exercise Questionnaire (BREQ) measures the stages of the self-determination contin. Subscales: Amotivation, External regulation, Introjected regulation, Identified regulation, Integrated regulation, Intrinsic regulation.Greater scores (averaged of outcome of respective subscale/items) indicate greater tendency for exercise behaviour to be regulated by particular construct (respective subscale).
Self-reported assessment of motivation to eat healthily | Assessed at start of study - through study completion - up to 4-5 weeks
  To examine the influence of self-reported motivation to adopt healthy eating behaviour on the relationship between experimental conditions and study outcomes. Scale involve:
  Regulation of Eating Behavioural Scale (REBS). Subscales: Amotivation, External regulation, Introjected regulation, Identified regulation, Integrated regulation, Intrinsic regulation. Greater scores (averaged of outcome of respective subscale/items) indicate greater tendency for eating behaviour to be regulated by particular construct (respective subscale).
Self-reported attitudes towards eating behaviour as assessed by the Three Factor Eating Behaviour Questionnaire (TFEQ-R18) | Assessed at start of study - through study completion - up to 4-5 weeks
  Influence of self-reported attitudes towards eating on the relationship between experimental conditions and study outcomes. Scale involve:
  Three Factor Eating Behaviour Questionnaire (TFEQ-R18) Subscales: Dietary Restraint, Uncontrolled Eating, Emotional Eating Greater scores (averaged outcome of respective subscale/items) indicate greater likelihood of the behaviour (of construct measure by respective subscales).
Self-reported weight-related behaviour change status as assessed by the Physical Activity Stages of Change Questionnaire | Assessed at start of study - through study completion - up to 4-5 weeks
  Influence of self-reported weight-related behaviour change status on the relationship between experimental conditions and study outcomes. Scale involve:
  Physical Activity Stages of Change Questionnaire. Scores (based on scoring algorithm) will indicate participants' current stage of motivational readiness for change specific to physical activity. Greater score (1-5 representing five stages of change) indicates physical activity status and intent to be active.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF)
  Will be made available to other researchers upon request